CLINICAL TRIAL: NCT03528850
Title: Stony Brook Telehealth Study. Tele-transitions of Care. An Approach to Reduce 30-day Readmission Using Tele-Health Technology; A Randomized Controlled Trial
Brief Title: Stony Brook Telehealth Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 970227
Record Dates: First submitted 2018-02-01; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Telemedicine; Patient Readmission

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth (Experimental): The Telehealth arm will receive daily biometric measurement of blood pressure, heart rate, oxygen saturation and weight. The Telehealth arm will also have weekly virtual visits for the first month after hospital discharge. The Telehealth arm will answer surveys weekly for the first 30 days.
  Interventions: Other: Telemedicine evaluation
- Standard of Care (No Intervention): The Standard of Care will receive no interventions but will conduct surveys at enrollment and at the end of 30 days.

INTERVENTIONS:
Other: Telemedicine evaluation — Weekly virtual visits and daily biometric readings of blood pressure, weight, oxygen saturation and pulse
  Arms: Telehealth

SUMMARY:
The study evaluates the feasibility of providing tele-transition of care, using risk stratification, novel data tools, remote patient monitoring and virtual visits. A new communication tool for relaying tele-communication among providers caring for the virtual patient is introduced. The primary endpoint is 30-day readmissions.

DETAILED DESCRIPTION:
The objective is to evaluate the feasibility and effectiveness of a patient-centered, physician led, transition of care, telehealth intervention. The intervention begins at the bedside prior to hospital discharge and involves remote patient monitoring of daily vitals, weekly virtual visits, detailed Electronic Medical Record (EMR) documentation and use of risk stratification as well as data from the Health Information Exchange (HIE).

The hypothesis is that in comparison to standard care:

1. Preventable hospital readmissions will be reduced through patient-centered virtual visits, daily biometric surveillance, and increased data access.
2. Patient satisfaction during the transition of care period will be improved
3. Adverse healthcare outcomes leading to ED visits or death will be reduced The primary aim of the study is to determine the effect of telehealth on unplanned hospital readmissions within 30 days of the index hospitalization discharge. In addition, data is collected in order to provide secondary analyses on the effect of telehealth on emergency department utilization, patient satisfaction, qualitative patient experience, patient self-management and self-efficacy attitudes.

The Telehealth patient is provided with a smart phone device and Bluetooth-enabled blood pressure monitoring cuff, weighing scale, and pulse oximeter. Telehealth patients measure their vitals daily and have weekly virtual visits with a transition of care physician (teledoc). The teledoc in this trial, is a senior resident physician in preventive medicine or family medicine.

Patient enrollment and randomization occurs at the bedside prior to hospital discharge. All patients are consented for the HIE in addition to the trial, and are risk stratified though an EMR data, based validated algorithm. The care management team is notified of all study participants in order to communicate to the telehealth team the date and time of hospital discharge. An introduction is made in person with the teledoc to evaluate the patient in person prior to virtual visits. Upon hospital discharge the patient receives the telehealth equipment by a vendor service to their home within 48 hours.

Risk stratification is done by an internally and externally validated High Risk Readmission Tool across many different hospital systems.

The patient follows prompts from the smart phone to register vitals daily, using a blood pressure cuff, pulse oximeter and digital scale. The teledoc determines the safety range parameters of the vitals depending on the patient clinical history and status. The telehealth vendor, notifies the teledoc of any abnormal values.

Weekly telehealth visits are conducted for the first 30 days after a hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Family Medicine Patients who are:

  * Age 30 years or older
  * Able to provide consent for their own care
  * English speakers (able to comprehend and speak English)
  * Patients with good cognitive function (as evidence by ability to answer a mild cognitive screen (age, telephone, current date, name of facility)
  * Living within reasonable commute to the Family Medical Group clinics
  * Patients with a life expectancy greater than 6 months
  * Patients with a clinical disposition to home after hospital discharge
  * Patients that are able to turn on the telehealth technology and follow prompts

Exclusion Criteria:

* Uninsured patients who are not currently seen by the Family Medicine Practice
* Patients whose physical limitations prohibit the use of the telehealth equipment
* Patients involved in another research study
* Pregnant patients (patients actively trying to conceive)
* Admission for a psychiatric primary diagnosis

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Readmission | 30 Days
  Hospital Readmission is calculated by data abstracted from the Electronic Medical Record and by surveys. Study data is collected and managed using REDCap (16) electronic data capture tools hosted at Stony Brook Medicine. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources. REDCap software allows the team to incorporate a randomization schema to include it in the process of enrollment seamlessly. After meeting inclusion criteria, the software follows a schema unknown to the researchers to randomly select consented participants into appropriate arms of trial.

SECONDARY OUTCOMES:
Emergency Room Utilization | 30 Days
  Emergency Room Utilization is calculated by data abstracted from the Electronic Medical Record and by surveys. Study data is collected and managed using REDCap (16) electronic data capture tools hosted at Stony Brook Medicine. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources. REDCap software allows the team to incorporate a randomization schema to include it in the process of enrollment seamlessly. After meeting inclusion criteria, the software follows a schema unknown to the researchers to randomly select consented participants into appropriate arms of trial.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Noel, MD MPH, Study Director — Stony Brook Medicine Telehealth Director
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and supporting data will be shared with other similar academic centers upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available within 1 year of publication and will be available for 5 years.

REFERENCES:
- [Derived] Noel K, Messina C, Hou W, Schoenfeld E, Kelly G. Tele-transitions of care (TTOC): a 12-month, randomized controlled trial evaluating the use of Telehealth to achieve triple aim objectives. BMC Fam Pract. 2020 Feb 7;21(1):27. doi: 10.1186/s12875-020-1094-5. PMID 32033535